CLINICAL TRIAL: NCT06388187
Title: Efficacy and Safety of Cagrilintide s.c. in Combination With Semaglutide s.c.(CagriSema s.c. 1.0 mg/1.0 mg and 1.7 mg/1.7 mg) Once-weekly in Participants With Overweight or Obesity
Brief Title: A Research Study to See How Well Different Doses of CagriSema Help People With Excess Body Weight Lose Weight
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-7749; U1111-1298-3451 (Other: World Health Organization (WHO)); 2023-509273-24 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CagriSema Dose 1 (Experimental): Participants will receive once-weekly subcutaneous (s.c) injections of CagriSema (cagrilintide and semaglutide) at escalating doses every week in 8-week dose escalation period until target dose (dose 1) of CagriSema (cagrilintide and semaglutide) is achieved and maintained up to 60 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Placebo Dose 1 (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to cagrisema dose 1 (cagrilintide and semaglutide) for 68 weeks.
  Interventions: Drug: Placebo
- CagriSema Dose 2 (Active Comparator): Participants will receive once-weekly s.c injections of CagriSema (cagrilintide and semaglutide) at escalating doses every week in 12-week dose escalation period until target dose (dose 2) of CagriSema(cagrilintide and semaglutide) is achieved and maintained up to 56 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Placebo Dose 2 (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to cagrisema dose 2 (cagrilintide and semaglutide) for 68 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive once-weekly cagrilintide subcutaneously.
  Arms: CagriSema Dose 1; CagriSema Dose 2
Drug: Semaglutide — Participants will receive once-weekly semaglutide subcutaneously.
  Arms: CagriSema Dose 1; CagriSema Dose 2
Drug: Placebo — Participants will receive once-weekly placebo matched to cagrilintide and semaglutide subcutaneously.
  Arms: Placebo Dose 1; Placebo Dose 2

SUMMARY:
This study will look at how well CagriSema helps people with excess body weight lose weight. CagriSema is a new medicine developed by Novo Nordisk that combines cagrilintide and semaglutide. CagriSema cannot yet be prescribed by doctors. In the study, participant will either get CagriSema or dummy medicine and which treatment participant get is decided by chance. The study will last for about 1½ years for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age above or equal to 18 years at the time of signing informed consent

  1. Body Mass index (BMI) greater than or equal to (≥) 30.0 kilogram per meter square (kg/m^2) or
  2. BMI ≥27.0 kg/m2 with the presence of at least one obesity related complication including, but not limited to hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease

Exclusion Criteria:

* Glycated haemoglobin (HbA1c) ≥6.5% (48 millimoles per mole [mmol/mol]) as measured by the central laboratory at screening
* History of type 1 or type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-04-21 (Estimated); Study Completion 2026-04-21 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%).
Achievement of ≥5% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participant.

SECONDARY OUTCOMES:
Achievement of ≥10% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participant.
Achievement of ≥15% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participant.
Achievement of ≥20% weight reduction | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participant.
Change in waist circumference | From baseline (week 0) to end of treatment (week 68)
  Measured in centimeter (cm).
Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 68)
  Measured in millimeters of mercury.
Ratio to baseline in lipids: Total cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: High-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: Low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: Very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: Triglycerides | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Ratio to baseline in lipids: Free fatty acids | From baseline (week 0) to end of treatment (week 68)
  Measured in ratio.
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to end of study (week 74)
  Measured as count of events.
Number of treatment emergent serious adverse events (TESAEs) | From baseline (week 0) to end of study (week 74)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (25):
- United States (7):
  - Aurora FDRC Inc., Costa Mesa, California
  - Clinical Trial Res Assoc,Inc, Plantation, Florida
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - Accellacare, Wilmington, North Carolina
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Washington Cntr Weight Mgmt, Arlington, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
- Canada (3):
  - Ocean West Research Clinic, Surrey, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Wharton Med Clin Trials, Hamilton, Ontario
- France (4):
  - Hospices Civils de Lyon-Hopital Lyon Sud-1, Pierre-Bénite
  - Hospices Civils de Lyon-Hopital Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec, Saint-Herblain
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil, Toulouse
- Germany (5):
  - InnoDiab Forschung GmbH, Essen
  - Wendisch - Dahl Hamburg - DZHW, Hamburg
  - AmBeNet GmbH, Leipzig
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - Forschungszentrum Ruhr KliFoCenter GmbH, Kahrmann, Witten
- United Kingdom (6):
  - The Health Centre, Bradford-on-Avon
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital_Cambridge, Cambridge
  - University Hospital Coventry - WISDEM Centre, Coventry
  - Staploe Medical Centre, Soham
  - Joint Clinical Research Facility - Swansea, Swansea

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com